CLINICAL TRIAL: NCT02380872
Title: Cytokine (IL-1ß) and Matrix Metalloproteinase (MMP) Levels in Gingival Crevicular Fluid After Use of Platelet Rich Fibrin or Connective Tissue Graft in the Treatment of Localized Gingival Recessions
Brief Title: Cytokine and MMP Levels in Gingival Crevicular Fluid in the Treatment of Localized Gingival Recessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Gülnihal Eren, Research Asisstant, Research Assistant, Ege University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: Ege Uni School of Dentistry
Record Dates: First submitted 2015-02-14; First posted 2015-03-05 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Gingival Recession
Keywords: Gingival recession; fibrin; connective tissue; gingival crevicular fluid; matrix metalloproteinase; cytokine
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Connective tissue graft (Active Comparator): Connective tissue graft Soft tissue harvested from palatum of the subjects.
  Interventions: Procedure: Connective tissue graft
- Platelet Rich Fibrin (Experimental): Autogenous platelet and leukocyte fibrin material was obtained from blood.
  Interventions: Procedure: Platelet Rich Fibrin

INTERVENTIONS:
Procedure: Connective tissue graft — gingival recession treated with connective tissue graft
  Arms: Connective tissue graft
Procedure: Platelet Rich Fibrin — gingival recession treated with platelet rich fibrin
  Arms: Platelet Rich Fibrin

SUMMARY:
The main objective of this study was to evaluate the matrix metalloproteinase (MMP)-8, and -9, tissue inhibitor of matrix metalloproteinase and interleukin-1beta levels in gingival crevicular fluid during the early and late stages of healing for gingival recession sites treated by coronally advanced flap plus platelet rich fibrin (PRF) compared to CAF plus connective tissue graft. As PRF consists of several growth factors, it may enhance the healing potential of soft tissues, the investigators hypothesized that using PRF in the treatment of gingival recessions might regulate inflammation and promote wound healing.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effect of PRF by assessing gingival crevicular fluid (GCF) levels of MMP-8, MMP-9, tissue inhibitor of matrix metalloproteinase (TIMP-1) and interleukin-1beta (IL-1β) during the early and late stages of healing following coronally advanced flap (CAF) plus PRF or CAF plus connective tissue graft (CTG) treatment.

Primary outcome variables were biochemical parameters, such as: GCF MMP-8, -9, TIMP-1 and IL-1β levels. The secondary outcome variables were change in gingival recession expressed as recession reduction in millimeters at follow-up visits.

Sample size has been estimated in 24 subjects per treatment groups. Random allocation of the treatment sites to test (CAF+ PRF) and control (CAF + SCTG) groups will be performed using a computerized selection of random numbers for allocation of the study groups.

Biochemical parameters: GCF samples were obtained from each recession defect in each subject immediately prior to treatment of recessions and at 10 days, 1 month, 3 months and 6 months after surgery.

Periodontal parameters including probing depth (PD), clinical attachment level (CAL), and gingival recession parameters including recession depth (RD), recession width (RW), and keratinized tissue width (KTW),were assessed by a calibrated examiner. At baseline and at 6 months, PD, RD, RW and KTW were evaluated by clinical assessment.

Follow-up of subjects: 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Similar bilateral Miller Class I or II localized gingival recessions at least ≥ 2 mm located on incisors, canines or premolars on both jaws
* Identifiable cementoenamel junction
* Age ≥ 18 years
* Presence of tooth vitality and absence of restorations and superficial caries in the area to be treated
* No periodontal surgical treatment in the previous 24 months on the involved sites
* Sufficient palatal donor tissue for the indicated SCTG.

Exclusion Criteria:

* Smoking
* Patients with a pregnancy or lactation period or self-reported history of antibiotic medication within three months
* Molar, mobile or teeth with crown or filling were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-10; Primary Completion 2013-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in MMP-8 gingival crevicular fluid level at 10 days, 1, 3 and 6 months | Baseline, 10 days, 1, 3 and 6 months
Change from Baseline in MMP-9 gingival crevicular fluid level at 10 days, 1, 3 and 6 months | Baseline, 10 days, 1, 3 and 6 months
Change from Baseline in TIMP-1 gingival crevicular fluid level at 10 days, 1, 3 and 6 months | Baseline, 10 days, 1, 3 and 6 months
Change from Baseline in IL-1beta gingival crevicular fluid level at 10 days, 1, 3 and 6 months | Baseline, 10 days, 1, 3 and 6 months

SECONDARY OUTCOMES:
Gingival recession depth | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gülnihal Eren, PhD. Dr., Principal Investigator — Ege University School of Dentistry; Gül Atilla, Professor, Study Director — Ege University School of Dentistry
Locations (1):
- Ege University School of Dentistry Department of Periodontology, Izmir, Turkey (Türkiye)